CLINICAL TRIAL: NCT03443089
Title: Comparative Bioavailability Study of Two Injectable Suspension Formulations, a Test (Medroxyprogesterone Acetate 25 mg/mL + Estradiol Cypionate 5 mg/mL) vs. a Reference (Medroxyprogesterone Acetate 25 mg/AMP + Estradiol Cypionate 5 mg/AMP)
Brief Title: Comparative Bioavailability of Two Injectable Suspension Formulations of Medroxyprogesterone Acetate+Estradiol Cypionate
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Galeno Desenvolvimento de Pesquisas Clínicas (Other Government)
Collaborators: Biolab Sanus Farmaceutica (Industry)
Responsible Party: Principal Investigator, Gilberto De Nucci, Doctor, Galeno Desenvolvimento de Pesquisas Clínicas
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GDN 022/16
Record Dates: First submitted 2018-02-16; First posted 2018-02-22 (Actual); Last update posted 2018-02-23 (Actual); Status verified 2018-02

CONDITIONS: Contraception
Keywords: medroxyprogesterone acetate; estradiol cypionate; bioavailability; monthly contraceptive

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test formulation (Experimental): Single intramuscular dose administration (1 ampoule) of medroxyprogesterone acetate 25 mg/mL+ estradiol cypionate 5 mg/mL (Depomês®, Biolab Sanus Farmacêutica Ltda.)
  Interventions: Drug: Test formulation
- Reference formulation (Active Comparator): Single intramuscular dose administration (1 ampoule) of medroxyprogesterone acetate 25 mg/ampole + estradiol cypionate 5 mg/ampole (Cyclofemina®, Millet Roux Ltda.)
  Interventions: Drug: Reference formulation

INTERVENTIONS:
Drug: Test formulation — Administration of a single intramuscular dose of an injectable formulation containing medroxyprogesterone acetate 25 mg/mL + estradiol cypionate 5 mg/mL after an overnight fast.
  Arms: Test formulation
Drug: Reference formulation — Administration of a single intramuscular dose of an injectable formulation containing medroxyprogesterone acetate 25 mg/ampole + estradiol cypionate 5 mg/ampole after an overnight fast.
  Arms: Reference formulation

SUMMARY:
This clinical trial evaluated the comparative bioavailability of two injectable suspension formulations of medroxyprogesterone acetate + estradiol cypionate, a test (Depomês®, 25 mg/mL medroxyprogesterone acetate + 5 mg/mL estradiol cypionate, Biolab Sanus Farmacêutica Ltda.) and a reference formulation (Cyclofemina®, 25 mg/0.5 mL medroxyprogesterone acetate + 5 mg/0.5 mL estradiol cypionate, Millet Roux Ltda.) in healthy female volunteers after a single intramuscular dose administration. In addition, this study also evaluated the safety and tolerability of these drugs.

DETAILED DESCRIPTION:
This study was performed in a monocentric, open label, parallel design, with 2 treatments, 1 period, in which twelve subjects received the test product (Depomês®, 25 mg/mL medroxyprogesterone acetate + 5 mg/mL estradiol cypionate, Biolab Sanus Farmacêutica Ltda.) and twelve subjects received the reference product (Cyclofemina®, 25 mg/0.5 mL medroxyprogesterone acetate + 5 mg/0.5 mL estradiol cypionate, Millet Roux Ltda.). The formulations (test or reference) were administered in a single intramuscular dose (1 ampoule) after an overnight fast (approximately 8 h). Blood samples (9 mL) were collected via a venous catheter into heparinized tubes at times pre-dose (0 h) and 6, 12, 24, 48, 72, 96, 120, 168, 240, 288, 336, 432, 504, 672, 840, 1008, 1176, 1344, 1512, 1680, 1848, and 2016 h after drug administration to measure medroxyprogesterone; and pre-dose (-48, -24 and 0 h) e 2, 4, 6, 8, 10, 12, 24, 48, 72, 96, 120, 168, 240, 288, 336, 432, 504, 672, 840, and 1008 h after drug administration to measure estradiol cypionate.

The safety assessment was based on recording adverse events throughout the study duration. The subjects systolic and diastolic pressures, heart rate and temperature were determined prior and at approximately 4, 8 and 12 h after drug administration. The clinical evaluation and the laboratory tests were also performed at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Body-mass index (BMI) ≥19.0 kg/m² and ≤ 27.5 kg/m²
* With regular cycles, without use of hormonal contraceptives (pills at least 3 months and injectables at least 1 year) and not using hormone replacement therapy
* Not pregnant or breastfeeding
* Good state of health
* Non-smoker or ex-smoker for at least 6 month
* Written informed consent, after having been informed about benefits and potential risks of the clinical trial, as well as details of the insurance taken out to cover the subjects participating in the clinical trial

Exclusion Criteria:

* Existing cardiac, hepatic and/or haematological diseases or pathological findings, which might interfere with the safety or tolerability and/or pharmacokinetics and/or pharmacodynamics of the active ingredient
* History of relevant central nervous system (CNS) and/or psychiatric disorders and/or currently treated CNS and/or psychiatric disorders
* Known allergic reactions to the active ingredients used or to constituents of the pharmaceutical preparations
* Subjects with severe allergies or multiple drug allergies, unless it is judged as not relevant for the clinical trial by the investigator
* Positive anti-HIV-test (if positive to be verified by western blot), HBs-AGtest (if positive to be verified by test for HBc-IgM) or anti-HCV-test
* Admitted for any reason up to 8 weeks before the start of the first treatment period of this study
* History of or current drug or alcohol dependence
* Subjects who are on a diet which could affect the pharmacokinetics of the active ingredient
* Regular intake of caffeine containing food or beverages of ≥ 500 mg caffeine per day
* Blood donation or other blood loss of more than 400 ml within the last 3 months prior to individual enrolment of the subject
* Participation in a clinical trial during the last 6 months prior to individual enrolment of the subject
* Positive pregnancy test, delivery or abortion in the 12 weeks prior to the planned hospitalization date.
* Subjects who are unable to understand the written and verbal instructions, in particular regarding the risks and inconveniences they will be exposed to during their participation in the clinical trial

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2017-03-31 (Actual); Primary Completion 2017-04-02 (Actual); Study Completion 2017-08-01 (Actual)

PRIMARY OUTCOMES:
Measurement of medroxyprogesterone acetate and estradiol cypionate plasma levels | 0-1008 hours after drug administration
  Blood sampling for the determination of plasma levels of medroxyprogesterone acetate and estradiol cypionate in participants of each treatment group.
Measurement of estradiol cypionate plasma levels | -48 to 1008 hours after drug administration
  Blood sampling for the determination of plasma levels of estradiol cypionate in participants of each treatment group.

SECONDARY OUTCOMES:
Maximum Plasma Concentration (Cmax) of medroxyprogesterone acetate | 0 - 1008 hours after drug administration
  Determination of maximum plasma concentration of medroxyprogesterone acetate on plasma concentrations of samples obtained.
Maximum Plasma Concentration (Cmax) of estradiol cypionate | 0 - 1008 hours after drug administration
  Determination of maximum plasma concentration of estradiol cypionate on plasma concentrations of samples obtained.
Area Under the Curve (AUC) of medroxyprogesterone acetate | 0 - 1008 hours after drug administration
  Determination of area Under the Curve of medroxyprogesterone acetate from plasma concentrations versus time curve of samples obtained.
Area Under the Curve (AUC) of estradiol cypionate | 0 - 1008 hours after drug administration
  Determination of area Under the Curve of estradiol cypionate from plasma concentrations versus time curves of samples obtained.
Number of adverse events per participant | Up to 1008 hours after drug administration
  Number of adverse events, in each treatment group, including clinically relevant alterations of vital signs and laboratory tests results.

CONTACTS AND LOCATIONS:
Overall Officials: Gilberto De Nucci, Doctor, Principal Investigator — Galeno Desenvolvimento de Pesquisas Clinicas Ltda
Locations (1):
- Galeno Desenvolvimento de Pesquisas Clinicas Ltda. - ME, Campinas, São Paulo, Brazil